CLINICAL TRIAL: NCT05607303
Title: Effect of Hormones on Frequency of Headache and Brain Structure and Function in Puberty
Status: Active, not recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20-1824
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Headache; Gender Identity
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: MTF youth who will begin taking estrogen clinically in < 6 months with or without headache
  Interventions: Other: Clinical estrogen therapy
- Controls: Cisgender males with or without headache

INTERVENTIONS:
Other: Clinical estrogen therapy — No research interventions will be used as a part of the study since the research is observational. Estrogen treatment will be prescribed and followed by participant's clinical physician.
  Groups: Cases

SUMMARY:
With a rising population of transgender adults and youth, there is a need for more research to meet the needs of this community. Transfemale (MTF) youth (male sex, female gender identity) who begin clinical Gender Affirming Hormone Therapy (GAHT) with estrogen may be at a higher risk for headache since estrogen has been linked to headache in cisgender females (female sex, female gender identity). This research hopes to learn more about headache in MTF youth.

DETAILED DESCRIPTION:
MTF youth who will begin estrogen clinically will be enrolled in the study and will be seen twice, once before starting estrogen and then one year after beginning estrogen. Cisgender males (male sex, male gender identity) will also be enrolled as a control group and will be seen once at the beginning of the study and then once a year later. The researchers will track how often youth have headaches during this time to see if it is different between groups. In a subset of the youth enrolled, an MRI will be completed to also look at brain structure and function.

ELIGIBILITY:
Inclusion Criteria:

For MTF youth (cases):

* Identify as MTF
* Age 11-20 years at the time of enrollment
* Plan to start estrogen clinically in < 6 months

For cisgender male youth (controls):

* Identify as cisgender male
* Age 9-20 years at the time of enrollment
* No diagnosis of Klinefelter Syndrome (XXY)

Exclusion Criteria:

* Cognitive, or psychiatric impairment resulting in inability to tolerate the study procedures not including depression or anxiety
* Known history of stroke, multiple sclerosis, or other serious neurologic condition

  * MRI-specific exclusion criteria (Weight > 500 lbs, claustrophobia, metal in body)

Ages: 9 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Transfemale (MTF) youth (male sex, female gender identity) and cisgender males (male sex, male gender identity) will be recruited for the study.
Study Population: Study population is limited to transgender females (male sex, female gender identity) for the case population and cisgender males (male sex, male gender identity) for the purposes of the study analysis as outlined in the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in frequency of headache. | 1 year
  Measured by headache count from daily headache diary.

SECONDARY OUTCOMES:
Change in amygdala structure. | 1 year
  Amygdala volume as measured on MRI.
Change in resting state functional connectivity pattern. | 1 year
  Measured by proportion of between-module connectivity patterns vs. within-module connectivity patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hranilovich, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No